CLINICAL TRIAL: NCT02826629
Title: "MADOCS: Manual Dexterity and Oculomotor Control as Vulnerability Markers in Schizophrenia"
Brief Title: "Manual Dexterity and Oculomotor Control in Schizophrenia"
Acronym: MADOCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier St Anne (Other)
Collaborators: University of Paris 5 - Rene Descartes (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D16-P01
Record Dates: First submitted 2016-05-20; First posted 2016-07-11 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Schizophrenia
Keywords: Sensorimotor Integration; Schizophrenia; TMS; Oculomotor; Motor Control
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Schizophrenia (Other): 40 patients with diagnosis of schizophrenia (25 medicated - 15 non-medicated)
  Interventions: Device: Manual dexterity; Device: Oculomotor movements; Device: TMS coupled to EMG recording; Other: Psychopathological evaluations; Other: Neuropsychological evaluations
- Healthy sibling (Other): 25 healthy siblings
  Interventions: Device: Manual dexterity; Device: Oculomotor movements; Device: TMS coupled to EMG recording; Other: Psychopathological evaluations; Other: Neuropsychological evaluations
- Ultra high risk for developing Schizophrenia (Other): 15 patients with ultra high risk for developing Schizophrenia
  Interventions: Device: Manual dexterity; Device: Oculomotor movements; Device: TMS coupled to EMG recording; Other: Psychopathological evaluations; Other: Neuropsychological evaluations
- Controls (Other): -25 age and gender-matched healthy controls
  Interventions: Device: Manual dexterity; Device: Oculomotor movements; Device: TMS coupled to EMG recording; Other: Psychopathological evaluations; Other: Neuropsychological evaluations

INTERVENTIONS:
Device: Manual dexterity — Control of manual dexterity will be assessed by a force sensor (Power Grip Manipulandum, PGM)
Device: Oculomotor movements — Oculomotor movements during behavioral task will be recorded using a video-oculography device
Device: TMS coupled to EMG recording — The involvement of cortical inhibition in this volitional inhibition task will be studied by neuronavigation guided TMS coupled to EMG recording
Other: Psychopathological evaluations
Other: Neuropsychological evaluations

SUMMARY:
The investigators recently showed that visuomotor integration was significantly altered in schizophrenic patients during: (i) a grip force task (Teremetz et al., 2014), and (ii) a saccadic paradigm (oculomotor task)(Amado et al., 2008). Given this findings, the investigators propose a combined study of oculomotor and grip force control to better characterize the sensorimotor integration deficit. This approach may allow for identification of behavioural biomarkers of vulnerability to develop schizophrenia.

DETAILED DESCRIPTION:
1 - Scientific background and rational Use of sensory cues is essential for execution and correction of voluntary movements. The motor areas and their regulation is of special interest in patients with schizophrenia as there is clear evidence of motor abnormalities independent of the effects of antipsychotic medication, even before the onset of the disorder. Sensorimotor abnormalities have been proposed as a valid endophenotype in schizophrenia. Our global objective is to study and provide vulnerability markers for schizophrenia.

1. Control of manual dexterity will be assessed by a force sensor (Power Grip Manipulandum, PGM)
2. Oculomotor movements during behavioral task will be recorded using a video-oculography device
3. The involvement of cortical inhibition in this volitional inhibition task will be studied by neuronavigation guided TMS coupled to EMG recording

2 - Description of the project methodology There is strong evidence for schizophrenia being a neuro-developmental disorder (Rapoport et al., 2005). It has been shown, for many years, that patients with schizophrenia exhibit abnormal patterns of sensorimotor integration (Manschreck et al., 1982), which is the capacity to integrate different sensory stimuli into appropriate motor actions. It is clinically relevant, in terms of early diagnosis and prevention, whether deficient sensorimotor integration is present in the prodromal phase of schizophrenia, and whether this constitutes a vulnerability marker for the disease.

Our global objective is to study the interactions and related substratum of oculomotor movements during force control task.

The secondary objectives:

(i) To show that increased motor noise is indeed present in schizophrenia. (ii) To show by TMS that cortical excitability in the primary motor cortex (M1) is task-modulated and decreased in schizophrenia.

(iii) Assess the role of deficient cortical inhibition in these behavioral deficits To this end, three different groups of subjects will be studied: schizophrenic patients, non-affected siblings, ultra high risk patients, non-treated schizophrenic patients and healthy control subjects.

ELIGIBILITY:
Inclusion Criteria:

* All groups:

  1. 18>yrs<50
  2. Medical visit completed
  3. Visual acuity (9/10 for each eye or corrected)
  4. Provided written informed consent
* Group of patient suffering from schizophrenia:

  4. DSM-IV-TR diagnostic criteria for schizophrenia 5. Treatment: stable atypical anti-psychotic medication for >3 months prior to the study
* Group of UHR patient:

  6. 18>yrs<30 7. Fulfill at risk criteria of CAARMS diagnostic tool

Exclusion Criteria:

• All groups:

1. IQ<70,
2. Contraindications for TMS protocol: no previous history of neurosurgery or seizures or 1st degree relative with history of seizures, heart disease, drug abuse or addiction in the last 12 months, medications that lower seizure threshold including clozapine, bupropion, méthadone or theophylline.
3. Metallic implant in head (except dental fillings)
4. Pacemaker, or other electronic implanted devices
5. Central neurological disease: parkinsonism, x
6. Severe heart attack
7. Instable clinical state (e.g. stroke)
8. Previous history of drug abuse lasting more than 5 years or during the last year
9. Life event with a moderate to severe impact
10. Caffeine intake in the last two hours preceding visuomotor assessment

    • Groups of Siblings and Healthy controls:
11. No previous history of psychiatric disease, psychotic spectrum disorder (according to DIGS 3.0)
12. No previous history of antipsychotic medication (entire life)

    • Groups of UHR patient:
13. Chlorpromazine dose >100mg over more than 12 weeks
14. No previous history of autism spectrum disorder, bipolar disorder or diagnozed schizophrenia (according to DSM-IV-TR criteria), isolated anxiety disorders (e.g. social phobia, agoraphobia)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2016-07-26 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Behavioural assessment | BASELINE
  Index reflecting motor performance during visuomotor task (including force and oculomotor control)

SECONDARY OUTCOMES:
Clinical scale : PANSS | BASELINE
  Positive and Negative Syndrome Scale: Assess positive and negative symptoms
Clinical scale : DIGS III | BASELINE
  Diagnostic Interview for Genetic Studies 3.0: Overview of clinical state
Clinical scale : BPRS | BASELINE
  Brief Psychiatric Rating Scale: Assess schizophrenic symptoms
Clinical scale : SAS | BASELINE
  Simpson Angus Extra-Pyramidal Scale: Asses extra-pyramidal signs
Clinical scale : AIMS | BASELINE
  Abnormal Involuntary Movements Scale: Assess abnormal involuntary movements
Clinical scale : TAP | BASELINE
  Test battery for Attentional Performance: Assess attentional capacity (e.g. working memory)
Clinical scale : Stroop | BASELINE
  Stroop color naming test: Assess selective attention or inhibition.
Clinical scale : WASI | BASELINE
  Wechsler Abbreviated Scale of Intelligence: Assess intelligence quotient
Tracking performance (motor task): RMS Error | BASELINE
  RMS Error (Root Mean Square)
Tracking performance (motor task): Coefficient of variability | BASELINE
  Coefficient of variability
Tracking performance (motor task): Timing | BASELINE
  Timing/inhibition
Ocolomotor performance (eye tracker) : Saccade | BASELINE
  Saccade error (back up/ catch up saccades) during smooth pursuit and fixation
Ocolomotor performance (eye tracker): Gain | BASELINE
  Gain (target velocity/gaze velocity), Reaction time
Ocolomotor performance (eye tracker): Amplitude of eye movements | BASELINE
  Amplitude (°) and velocity (°/s) of saccadic movements
Motor noise | BASELINE
  Variability of EMG response during visuomotor task
Cortical excitability (MEP; TMS) | BASELINE
  Motor evoked potential (MEP) during visuomotor task (single pulse TMS)
Cortical inhibition (SICI; TMS) | BASELINE
  Cortical inhibition measured during visuomotor task (paired-pulse TMS; MEP)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Amado, Dr, Study Director — CHSA; Pavel Lindberg, PhD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (2):
- France (2):
  - Centre de Recherche Clinique (CRC) - CHSA, Paris
  - Service Hospitalo-Universitaire (SHU) - CHSA, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Teremetz M, Amado I, Bendjemaa N, Krebs MO, Lindberg PG, Maier MA. Deficient grip force control in schizophrenia: behavioral and modeling evidence for altered motor inhibition and motor noise. PLoS One. 2014 Nov 4;9(11):e111853. doi: 10.1371/journal.pone.0111853. eCollection 2014. PMID 25369465
- [Background] Amado I, Landgraf S, Bourdel MC, Leonardi S, Krebs MO. Predictive saccades are impaired in biological nonpsychotic siblings of schizophrenia patients. J Psychiatry Neurosci. 2008 Jan;33(1):17-22. PMID 18197268